CLINICAL TRIAL: NCT02534038
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Efficacy of AVP-786 for the Treatment of Disinhibition in Patients With Neurodegenerative Disorders
Brief Title: Safety, Tolerability and Efficacy of AVP-786 for the Treatment of Disinhibition
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely because of difficulty with recruiting.
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-AVP-786-203
Record Dates: First submitted 2015-08-11; First posted 2015-08-27 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Disinhibition Syndrome
Keywords: Disinhibition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo drug to be taken twice a day for 6 weeks
  Interventions: Drug: Placebo
- AVP-786 (Active Comparator): Participants randomized to AVP-786 will take one dose of AVP-786 once a day and one dose of placebo once a day for the first 7 days; from day 8, participants will receive AVP-786 twice a day for 5 weeks.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786 — d6-DM/Q
  Other Names: Deuterated (d6)-dextromethorphan (DM)/Quinidine (Q)
  Arms: AVP-786
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
Treatment of disinhibition syndrome in participants with Neurodegenerative Disorder.

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of Neurodegenerative Disorder and must exhibit disinhibition syndrome of sufficient severity to warrant treatment.

This is a multicenter, randomized, double-blind, placebo-controlled, cross-over study consisting of two 6-week treatment periods.

Approximately 12 participants will be enrolled at approximately 2 centers in the United States.

Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of a Neurodegenerative Disorder including frontotemporal dementia, Alzheimer's disease (AD), progressive supranuclear palsy (PSP), corticobasal degeneration (CBD), dementia with Lewy bodies (DBL), vascular cognitive disorders, or Huntington's disease, at least 3 months prior to Baseline
* The participant has behavior from 2 of the 3 categories of disinhibited behavior from the definition of the behavioral variant of frontotemporal dementia
* The behavioral changes are not due to a pre-existing major psychiatric disorder (e.g., schizophrenia, bipolar disease, etc.) and are not due to the direct effect of systemic illness, drug action, or substance use
* Disinhibition scale score of ≥4 on the 3 core disinhibition items of the Frontal Behavioral Inventory (FBI) at Screening and Baseline

Exclusion Criteria:

* Participants with symptoms of disinhibition that is not secondary to Neurodegenerative Disorders
* Participants with myasthenia gravis
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy [except skin basal-cell carcinoma or untreated prostate cancer], poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AVP-786; Placebo: In Period 1, participants were randomized to receive AVP-786 (deuterated [d6]-dextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q]) once a day (OD) in the morning and placebo in the evening for the first 7 days of the study. From Day 8, participants received AVP-786 twice a day (BID) for 14 days. From Day 22, participants received a target dose of d6-DM 28 milligrams (mg)/Q 4.9 mg (AVP-786-28/4.9) BID for the remaining 3 weeks of Period 1. In Period 2, participants were randomized to receive matching placebo. The periods were separated by a 2-week washout period.
- Placebo; AVP-786: In Period 1, participants were randomized to receive matching placebo. In Period 2, participants were randomized to receive AVP-786 OD in the morning and placebo in the evening for the first 7 days of the study. From Day 8, participants received AVP-786 BID for 14 days. From Day 22, participants received a target dose of AVP-786-28/4.9 BID for the remaining 3 weeks of Period 2. The periods were separated by a 2-week washout period.
Period: Period 1 (6 Weeks)
Arm/Group | AVP-786; Placebo | Placebo; AVP-786
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Period 2 (6 Weeks)
Arm/Group | AVP-786; Placebo | Placebo; AVP-786
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A limited number of participants were enrolled prior to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | AVP-786; Placebo | Placebo; AVP-786 | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Reporting demographic data for this study in which only 1 participant was enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. |  | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Disinhibition Domain of the Neuropsychiatric Inventory (NPI)
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: No efficacy analyses were conducted due to the limited number of participants enrolled prior to study termination (N=1). In order to protect the privacy of participants, the results of enrolled participants cannot be reported.
Groups:
- Placebo: Participants received matching placebo in either the first or last 6 weeks of the study.
- AVP-786: Participants received up to a target dose of deuterated (d6)-dextromethorphan hydrobromide (d6-DM) 28 milligrams (mg)/quinidine sulfate (Q) 4.9 mg (AVP-786-28/4.9) twice a day (BID) in either the first or last 6 weeks of the study.
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline for the Total NPI Score
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Groups:
- AVP-786: Participants received up to a target dose of AVP-786-28/4.9 BID in either the first or last 6 weeks of the study.
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline for the NPI Total Caregiver Distress
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline for the NPI Disinhibition Domain Caregiver Distress
Time Frame: Baseline; Week 1, Week 3, Week 6, Week 8, Week 9, Week 11, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline for the Frontal Behavioral Inventory (FBI) Total Score
Time Frame: Baseline; Week 1, Week 3, Week 6, Week 8, Week 9, Week 11, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline for the FBI Disinhibition Domain Score
Time Frame: Baseline; Week 1, Week 3, Week 6, Week 9, Week 11, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From the First Assessment for the Modified Clinical Global Impression of Change (mCGIC) Scale
Time Frame: Week 3, Week 6, Week 11, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From the First Assessment for the Patient Global Impression of Change (PGIC) Scale
Time Frame: Week 3, Week 6, Week 11, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline for the Quality of Relationships (QoR) Scale
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline for the Quality of Life (QoL) Scale
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline for the Interpersonal Reactivity Index (IRI)
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline for the Center for Neurologic Study-Lability Scale (CNS-LS)
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline for the Mini-Mental State Examination (MMSE)
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline for the Cornell Scale for Depression in Dementia (CSDD)
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline for the Stroop Color and Word Task
Time Frame: Baseline; Week 6, Week 8, and Week 14
Population: as for outcome 1
Arm/Group | Placebo | AVP-786
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 22 weeks
Groups:
- Placebo: Participants received matching placebo for 6 weeks.
- AVP-786: Participants received AVP-786 (up to a target dose of d6-DM 28 milligrams [mg]/Q 4.9 mg [AVP-786-28/4.9] twice a day [BID]) for 6 weeks.
Arm/Group | Placebo | AVP-786
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | AVP-786 (N=1)
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02534038/Prot_SAP_000.pdf